CLINICAL TRIAL: NCT05869396
Title: Preoperative Echocardiography in Patients With Hip Fracture: A Prospective Cohort Study
Brief Title: Preoperative Echocardiography in Patients With Hip Fracture
Status: Completed | Type: Observational
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Carlo Rostagno, Asssociate Professor, University of Florence
Other Study IDs: CRostagno
Record Dates: First submitted 2023-04-25; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Perioperative Medicine; Hip Fractures; Echocardiography
Keywords: Elderly; Hip fracture; Prognosis; Echocardiography
MeSH Terms: conditions — Hip Fractures | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- echocardiogrpahy: Patients with with previously unknown systolic murmurs, unstable cardiovascular clinical conditions, recent (within 6 months) de-compensation of heart failure or hospital admission for coronary disease (high-risk group).
  Interventions: Diagnostic Test: echocardiography
- non echocardiography: Patients without previously unknown systolic murmurs, unstable cardiovascular clinical conditions, recent (within 6 months) de-compensation of heart failure or hospital admission for coronary disease (low-risk group).

INTERVENTIONS:
Diagnostic Test: echocardiography — Bedside echocardiography
  Groups: echocardiogrpahy

SUMMARY:
Aim of the study was to assess whether preoperative echocardiography affects time to surgery, length of hospital stay and in hospital mortality in patients undergoing hip fracture surgery. In the study entered two hundred fifty -five consecutive patients with hip fracture referred to a multidisciplinary hip fracture unit at a tertiary teaching hospital. Other 717 patients referred before implementation of routine echocardiographic examination were considered as control group. Echocardiography was performed in patients with systolic murmurs, unstable clinical conditions, recent decompensation of heart failure or hospital admission for coronary disease. Time to surgery, length of hospital stay (LOS) and in hospital mortality in patients underwent preoperative echocardiography (high risk group) were compared with patients who did not undergo echo (low-risk group ) and with an historical group.

DETAILED DESCRIPTION:
The study is part of a project of Italian Health Ministry and Toscana Region -Regional Fund -2010-2316600- and was approved by Ethical Committee of Regione Toscana. Written informed consent to treatment and collection of clinical data for research purposes was obtained at admission. The study, was conducted according to STROBE statements and performed in line with the principles of the Declaration of Helsinki.

Between Jan 1 and May 31 2018 255 consecutive patients with hip fracture aged > 70 years were referred to the Hip fracture Unit of a teaching hospital . The diagnosis of hip fracture was made according to Orthopaedic Trauma Association classification . All patients were evaluated by multidisciplinary hip fracture team according to a previously described protocol. Demographic data, comorbidities and functional status before trauma were recorded. According to local evaluation protocol echocardiography was performed in patients with previously unknown systolic murmurs, unstable cardiovascular clinical conditions, recent (within 6 months) decompensation of heart failure or hospital admission for coronary disease (high-risk group). Results were compared with patients without these characteristics, in whom echocardiography was not performed (low-risk group). Patients referred to hip fracture Unit in 2016 before implementation of echocardiography protocol were considered as control group.

ELIGIBILITY:
Inclusion Criteria:

* hip fragility fracture,
* age > 70 years

Exclusion Criteria:

* high energy fracture in aged > 70 years
* age < 70 years

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged > 70 years with hip fragility fracture
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 1 year]
  Mortality

SECONDARY OUTCOMES:
Relation between echocardiographic findings and survival | through study completion, an average of 1 year]
  Relation between echocardiographic findings and survival

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Rostagno, MD,PhD, Principal Investigator — University of Florence
Locations (1):
- UFlorence, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cartei A, Mossello E, Ceccofiglio A, Rubbieri G, Polidori G, Ranalli C, Cammilli A, Curcio M, Cavallini MC, Mannarino GM, Ungar A, Toccafondi G, Peris A, Marchionni N, Rostagno C. Independent, Differential Effects of Delirium on Disability and Mortality Risk After Hip Fracture. J Am Med Dir Assoc. 2022 Apr;23(4):654-659.e1. doi: 10.1016/j.jamda.2021.10.021. Epub 2021 Nov 30. PMID 34861226
- [Background] Rostagno C, Cartei A, Polidori G, Civinini R, Ceccofiglio A, Rubbieri G, Curcio M, Boccaccini A, Peris A, Prisco D. Management of ongoing direct anticoagulant treatment in patients with hip fracture. Sci Rep. 2021 May 4;11(1):9467. doi: 10.1038/s41598-021-89077-8. PMID 33947928
- [Result] Rostagno C, Cartei A, Rubbieri G, Ceccofiglio A, Civinini R, Curcio M, Polidori G, Boccaccini A. Hip Fracture Surgery in Severe Aortic Stenosis: A Study of Factors Affecting Mortality. Clin Interv Aging. 2022 Aug 4;17:1163-1171. doi: 10.2147/CIA.S360538. eCollection 2022. PMID 35957924